CLINICAL TRIAL: NCT01589874
Title: Anemia of Inflammation: Investigation on Impaired Iron Regulation in Acutely Ill Patients and Their Clinical Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: University of Milano Bicocca (Other)
Other Study IDs: 328/2007
Record Dates: First submitted 2012-03-06; First posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Anemia of Acute Inflammation
Keywords: hepcidin; anemia; acute inflammation; IL-6; cytokines
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, buffy coat
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- acute ill patients

SUMMARY:
Anemia of inflammation (AI), a normochromic, normocytic anemia, associated with abnormal iron utilization, erythropoietin hyporesponsiveness, and decreased red blood cells (RBC) survival is a very common problem in hospitalized patients for acute inflammatory diseases and develops within few days from the onset of illness. Deleterious effects of anemia include increased risk of cardiac related morbidity and mortality in critically ill and older patients.

Anemia is mediated by hepcidin, the 25-amino acid polypeptide hormone that is central to iron trafficking.

Several studies have been performed on pathophysiology of AI in patients affected by chronic diseases but few explore iron metabolism in humans with acute inflammation.

The aim is to develop effective new strategies to detect and manage AI in the setting of acutely ill patients, based on the understanding of iron balance underlying this disorder.

ELIGIBILITY:
Inclusion Criteria (both):

* serum C-reactive protein level > 3mg/dL
* creatinine level < 2mg/dL (clearance > 30%)

Exclusion Criteria:

* any haematological diseases
* cancer under chemotherapy
* AIDS (or HIV+)
* liver cirrhosis
* genetic hemochromatosis
* immunosuppressive therapy
* blood transfusion in the past 30-days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive patients admitted to Internal Medicine ward because of acute inflammatory illness
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-03 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
impact of acute inflammatory state on hemoglobin levels | 6 days - 8 days
  Hemoglobin levels, Blood Red Cells markers, C-RP and other routinary inflammatory markers on day 1 and day 6 (or 8), IL-1, IL-4, IL-6, IL-10, alpha-TNF, gamma-IFN, GDF-15, erythropoietin and hepcidin on day 1 and on day 6 (or 8)

SECONDARY OUTCOMES:
impact of acute inflammatory cytokines on hepcidin-driven iron balance and monocytes role in anemia of acute inflammation | 6 days - 8 days
  serum iron levels, ferritin and transferrin saturation, circulating monocytes and their HAMP mRNA.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Fabio, MD, PhD, Principal Investigator — Universita' degli Studi di Milano & Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico; Giovanna Fabio, MD, PhD, Study Director — Universita' degli Studi di Milano & Fondazione IRCCS Ca' Granda Osepdale Maggiore Policlinico
Locations (1):
- Internal Medicine Department - U.O. Medicina Interna 1/A, Via Francesco Sforza 35, Milan, Italy